CLINICAL TRIAL: NCT00792636
Title: Assessment of the Effect of Sumatriptan and Naproxen Sodium Combination Tablet, Sumatriptan Tablet, and Naproxen Sodium Tablet Treatment on Blood Pressure When Administered Intermittently for Six Months for the Acute Treatment of Migraine Attacks, With or Without Aura, in Adults
Brief Title: A Study to Determine the Effect of Sumatriptan and Naproxen Sodium Combination Tablet, Sumatriptan Tablet, and Naproxen Sodium Tablet on Blood Pressure When Treating Migraine Headaches That Occur During a 6-month Period
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110948
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Migraine Disorders
Keywords: sumatriptan and naproxen sodium; migraine with or without aura; naproxen sodium; sumatriptan; blood pressure; migraine headaches
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- sumatriptan and naproxen sodium combination (Experimental)
  Interventions: Drug: sumatriptan and naproxen sodium combination tablet
- sumatriptan (Active Comparator)
  Interventions: Drug: sumatriptan tablet
- naproxen sodium (Active Comparator)
  Interventions: Drug: naproxen sodium tablet

INTERVENTIONS:
Drug: sumatriptan and naproxen sodium combination tablet — sumatriptan 85mg and naproxen sodium 500mg
  Arms: sumatriptan and naproxen sodium combination
Drug: sumatriptan tablet — sumatriptan 85mg
  Arms: sumatriptan
Drug: naproxen sodium tablet — Naproxen sodium 500mg
  Arms: naproxen sodium

SUMMARY:
The purpose of this study is to test the effect on blood pressure of sumatriptan and naproxen sodium combination tablets, tablets containing only sumatriptan, and tablets containing only naproxen sodium when these drugs are taken to treat migraine headaches that occur during a 6-month period.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

* Male and female outpatients 18 to 65 years of age. Female subjects are eligible for participation in the study if they are:

  * Females of non-childbearing potential
  * Females of childbearing potential and who have a negative urine pregnancy test at Screening and agree to use one of the GlaxoSmithKline specified highly effective methods for avoiding pregnancy. Subjects taking oral contraceptives must be on a stable regimen for at least two months prior to Screening.
* Subject with migraines, with or without aura (ICHD-II criteria, 1.2.1 or 1.1) [International Headache Society, 2004]. Subject must have a history of two to eight attacks per month, on average, for the six months prior to the Screening Visit. Additionally the subject is to have experienced at least two, but no more than eight, migraine attacks per month for the three months prior to Screening Visit.
* Subject is able to distinguish migraine attacks from other headaches (i.e. tension-type headaches).
* Subject is willing and able to provide written informed consent, to comprehend and perform the requirements of the protocol.

Exclusion criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

* Subject has ≥10 migraine attacks or ≥15 headache days per month in total (including migraine, probable migraine or tension-type headache).
* Subject has retinal (ICHD-II 1.4), basilar (ICHD-II 1.2.6), or hemiplegic migraine (ICHD-II 1.2.4), or secondary headaches [International Headache Society, 2004].
* Subject has a history of controlled or uncontrolled hypertension or is currently taking any angiotension-converting enzyme (ACE) inhibitor or angiotension receptor blocker.
* Subject has an in-clinic screening blood pressure of ≥ 130/85 mmHg in two out of three blood pressure measurements.
* Subject is taking any anti-hypertensive medication for any reason including for migraine prophylaxis.
* Subject has a glycosylated hemoglobin ≥ 8.0
* Subject has a chronic condition (i.e. osteoarthritis, rheumatoid arthritis,fibromyalgia) which requires chronic daily administration of non-steroidal anti-inflammatory drugs (NSAIDS) (including acetaminophen) or opioids or opioid combination products.
* Subject, in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease.
* Subject has a history of congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in the study.
* Subject has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or any signs or symptoms consistent with any of the above.
* Subject has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold, or has been treated with an antiepileptic drug for seizure control within five years prior to Screening.
* Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in the study.
* Subject has hypersensitivity, allergy, intolerance or contraindication to the use of any triptan, NSAID, or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma.
* Subject is currently taking, or has used, an ergot or ergot-derived medication in the previous three months for migraine prophylaxis or is taking a medication that is not stabilized (i.e. change of a dose within the past two months) for chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized.
* Subject has a recent history of regular use of opioids or barbiturates for the treatment of their migraine headache and/or other non-migraine pain. Regular use is defined as an average of four days per month over the last six months.
* Subject has taken or plans to take a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum) or a CNS stimulant medication (such as atomoxetine, dextroamphetamine and amephetamine products, dexmethlyphenidate, lisdexamdetamine dimesylate and methylphenidate) anytime within two weeks prior to Screening through two-weeks post-treatment.
* Subject has a history of any bleeding disorder or is currently taking any anticoagulant or any anti-platelet agent. (except low-dose aspirin <=325mg/day for cardioprotective reasons).
* Subject has evidence or history of any gastrointestinal surgery, gastrointestinal ulceration or perforation in the past six months, gastrointestinal bleeding in the past year, or evidence or history of inflammatory bowel disease.
* Subject is pregnant, actively trying to become pregnant, or breast feeding or subject is not willing to have pregnancy tests performed as required.
* Subject tests positive for illicit substances on toxicology screen or has evidence of alcohol or substance abuse within the last year, or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
* Subject has participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (46):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Avon, Connecticut
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Harrisburg, North Carolina
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] White WB, Derosier FJ, Thompson AH, Adams BE, Goodman DK. Evaluation of the migraine treatment sumatriptan/naproxen sodium on blood pressure following long-term administration. J Clin Hypertens (Greenwich). 2011 Dec;13(12):910-6. doi: 10.1111/j.1751-7176.2011.00554.x. Epub 2011 Nov 11. PMID 22142350
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110948 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of participants defined as starting the study in the Participant Flow module includes only those participants randomized to treatment.
Groups:
- Sumatriptan/Naproxen: Sumatriptan 85 milligrams (mg) and naproxen sodium 500 mg combination tablet taken after migraine attack
- Sumatriptan: Sumatriptan 85 mg tablet taken after migraine attack
- Naproxen: Naproxen sodium 500 mg tablet taken after migraine attack
Period: Overall Study
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Started | 135 | 136 | 136
Completed | 67 | 55 | 55
Not Completed | 68 | 81 | 81
Not completed — Protocol Violation | 17 | 23 | 20
Not completed — Met Protocol-defined Stopping Criteria | 19 | 20 | 20
Not completed — Lost to Follow-up | 13 | 19 | 14
Not completed — Withdrew Consent | 10 | 13 | 9
Not completed — Lack of Efficacy | 3 | 4 | 13
Not completed — Adverse Event | 4 | 2 | 3
Not completed — Investigator Discretion | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen | Total
Number analyzed (Participants) | 122 | 112 | 118 | 352
Age, Continuous [Mean (Standard Deviation); unit: Years] — Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home blood pressure assessment. Not all randomized participants were part of the ITT Population.
  Years | 39.0 (11.64) | 39.8 (11.22) | 39.1 (11.92) | 39.3 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home blood pressure assessment. Not all randomized participants were part of the ITT Population.
  Participants
    Female | 94 | 98 | 96 | 288
    Male | 28 | 14 | 22 | 64
Race/Ethnicity, Customized [Number; unit: participants] — Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home blood pressure assessment. Not all participants were enrolled in the ITT Population.
  participants
    White | 108 | 96 | 105 | 309
    African American/African Heritage | 12 | 11 | 10 | 33
    Asian | 2 | 3 | 3 | 8
    Asian and White | 0 | 1 | 0 | 1
    American Indian or Alaska Native | 0 | 1 | 0 | 1
Average Number of Migraine Attacks per Month [Mean (Standard Deviation); unit: migraines] — Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home blood pressure assessment. The average number of migraines per month for the 6-month period prior to Screening is presented.
  migraines | 4.5 (1.76) | 4.2 (1.67) | 4.6 (1.8) | 4.4 (1.75)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan and Naproxen
Description: The calculation of baseline and post-baseline mean BP (either systolic or diastolic) for each month (30-day period) is the average of all valid Telephonic Self-Measured Blood Pressure (T-SMBP) measurements. T-SMBP technology is a method that allows the participant to self-measure BP outside the clinic using a BP monitor and transfer the data from their home to a central server. Change from baseline was calculated as the Month 6 value minus the Baseline value. Least squares mean and confidence intervals were based on mixed model repeated measures analysis (MMRM).
Time Frame: Baseline and Month 6
Population: ITT Population. Mean BP values were not available for all participants at baseline and Month 6 due to participant drop-out or to an inadequate number of BP collections.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sumatriptan | Naproxen
Number analyzed (Participants) | 109 | 115
mmHg
  Systolic, Baseline, n=109, 115 | 110.8 (9.15) | 110.1 (9.19)
  Systolic, Month 6, n=42, 37 | 109.4 (7.70) | 108.2 (9.16)
  Systolic, Change from Baseline, n=41, 36 | -2.8 (5.69) | -1.8 (6.53)
  Diastolic, Baseline, n=109, 115 | 75.7 (7.38) | 74.7 (7.00)
  Diastolic, Month 6, n=42, 37 | 73.9 (7.03) | 74.3 (8.47)
  Diastolic, Change from Baseline, n=41, 36 | -1.6 (4.21) | -0.6 (5.50)
Statistical Analysis 1: Comparison: Sumatriptan; Test type: Superiority or Other; Least-squares mean = -1.7, 95% CI 2-sided [-3.2 to -0.3] — Systolic Blood Pressure. The following covariates were used in this analysis: Age, Gender, Baseline migraines per month, Baseline blood pressure
Statistical Analysis 2: Comparison: Sumatriptan; Test type: Superiority or Other; Least-squares mean = -0.9, 95% CI 2-sided [-2.2 to 0.3] — Diastolic Blood Pressure. The following covariates were used in this analysis: Age, Gender, Baseline migraines per month, Baseline blood pressure
Statistical Analysis 3: Comparison: Naproxen; Test type: Superiority or Other; Least-squares mean = -1.9, 95% CI 2-sided [-3.4 to -0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Naproxen; Test type: Superiority or Other; Least-squares mean = -0.7, 95% CI 2-sided [-2.0 to 0.6] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan/Naproxen
Description: The calculation of baseline and post-baseline mean blood pressure (BP) (either systolic or diastolic) for each month (30-day period) is the average of all valid Telephonic Self-Measured Blood Pressure (T-SMBP) measurements. T-SMBP technology is a method that allows the participant to self-measure BP outside the clinic using a BP monitor and transfer the data from their home to a central server. Change from baseline was calculated as the Month 6 value minus the Baseline value. Least squares mean and confidence intervals were based on mixed model repeated measures analysis (MMRM).
Time Frame: Baseline and Month 6
Population: Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home BP assessment. Mean BP values were not available for all participants at baseline and Month 6 due to participant drop-out or to an inadequate number of BP collections.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Sumatriptan/Naproxen
Number analyzed (Participants) | 120
millimeters of mercury (mmHg)
  Systolic, Baseline, n=120 | 111.7 (9.00)
  Systolic, Month 6, n=48 | 107.1 (9.59)
  Systolic, Change from Baseline, n=47 | -2.9 (5.24)
  Diastolic, Baseline, n=120 | 76.0 (6.83)
  Diastolic, Month 6, n=48 | 73.0 (6.84)
  Diastolic, Change from Baseline, n=47 | -2.1 (4.44)
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen; Test type: Superiority or Other; Least-squares mean = -2.1, 95% CI 2-sided [-3.4 to -0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen; Test type: Superiority or Other; Least-squares mean = -1.5, 95% CI 2-sided [-2.6 to -0.3] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Treatment Difference in Systolic and Diastolic Blood Pressure Mean Changes From Baseline at 6 Months Between Sumatriptan/Naproxen and Sumatriptan
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Sumatriptan/Naproxen | Sumatriptan
Number analyzed (Participants) | 120 | 109
mmHg
  Systolic, Baseline, n=120, 109 | 111.7 (9.00) | 110.8 (9.15)
  Systolic, Month 6, n=48, 42 | 107.1 (9.59) | 109.4 (7.70)
  Systolic, Change from Baseline, n=47, 41 | -2.9 (5.24) | -2.8 (5.69)
  Diastolic, Baseline, n=120, 109 | 76.0 (6.83) | 75.7 (7.38)
  Diastolic, Month 6, n=48, 42 | 73.0 (6.84) | 73.9 (7.03)
  Diastolic, Change from Baseline, n=47, 41 | -2.1 (4.44) | -1.6 (4.21)
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Least-squares mean = 0.4, 95% CI 2-sided [-1.6 to 2.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Least-squares mean = 0.5, 95% CI 2-sided [-1.2 to 2.2] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Treatment Difference in Systolic and Diastolic Blood Pressure Mean Changes From Baseline at 6 Months Between Sumatriptan/Naproxen and Naproxen
Description: as for outcome 1
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sumatriptan/Naproxen | Naproxen
Number analyzed (Participants) | 120 | 115
mmHg
  Systolic, Baseline, n=120, 115 | 111.7 (9.00) | 110.1 (9.19)
  Systolic, Month 6, n=48, 37 | 107.1 (9.59) | 108.2 (9.16)
  Systolic, Change from Baseline, n=47, 36 | -2.9 (5.24) | -1.8 (6.53)
  Diastolic, Baseline, n=120, 115 | 76.0 (6.83) | 74.7 (7.00)
  Diastolic, Month 6, n=48, 37 | 73.0 (6.84) | 74.3 (8.47)
  Diastolic, Change from Baseline, n=47, 36 | -2.1 (4.44) | -0.6 (5.50)
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Least-squares mean = 0.3, 95% CI 2-sided [-1.7 to 2.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Least-squares mean = 0.8, 95% CI 2-sided [-0.9 to 2.5] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan/Naproxen for the ITT Subpopulation of Participants Treating, on Average, <4 Migraines, 4-6 Migraines, >=4 Migraines, and >6 Migraines Per Month
Description: The calculation of baseline and post-baseline mean BP (either systolic or diastolic) for each month (30-day period) is the average of all valid T-SMBP measurements. The subgrouping of the ITT population was created and examined to demonstrate the robustness of the results for the primary analysis.Descriptive statistics were calculated for baseline, month 6, and change from baseline to month 6. LSMeans and corresponding confidence intervals were based on MMRM analysis. LSMeans and corresponding confidence intervals were not calculated for > 6 migraines/month group due to lack of convergence.
Time Frame: Baseline and Month 6
Population: Intent-to-Treat (ITT) Population: all randomized participants who took at least one dose of investigational product and had at least one valid post-baseline at-home blood pressure assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sumatriptan/Naproxen
Number analyzed (Participants) | 122
mmHg
  Systolic, <4 migraines per month | -2.0 [-3.5 to -0.5]
  Systolic, 4-6 migraines per month | -3.3 [-7.0 to 0.4]
  Systolic, >=4 migraines per month | -3.7 [-6.7 to -0.7]
  Diastolic, <4 migraines per month | -1.2 [-2.5 to 0.00]
  Diastolic, 4-6 migraines per month | -5.3 [-9.9 to -0.6]
  Diastolic, >=4 migraines per month | -4.1 [-7.2 to -1.1]

6. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan/Naproxen for the ITT Subpopulation of Participants Treating, on Average, <1.3 Times Per Migraine, 1.3-1.7 Times Per Migraine, and >1.7 Times Per Migraine
Description: The calculation of baseline and post-baseline mean BP (either systolic or diastolic) for each month (30-day period) is the average of all valid T-SMBP measurements. The subgrouping of the ITT population was created and examined to demonstrate the robustness of the results for the primary analysis.Descriptive statistics were calculated for baseline, month 6, and change from baseline to month 6. LSMeans and corresponding confidence intervals were based on MMRM analysis.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sumatriptan/Naproxen
Number analyzed (Participants) | 122
mmHg
  Systolic, <1.3 doses per migraine | -0.3 [-2.7 to 2.0]
  Systolic, 1.3-1.7 doses per migraine | -2.7 [-5.3 to -0.2]
  Systolic, >1.7 doses per migraine | -3.8 [-6.2 to -1.5]
  Diastolic, <1.3 doses per migraine | -0.4 [-2.2 to 1.5]
  Diastolic, 1.3-1.7 doses per migraines | -0.9 [-2.9 to 1.2]
  Diastolic, >1.7 doses per migraine | -3.2 [-5.3 to -1.0]

7. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan/Naproxen for the ITT Subpopulation of Participants Treating, on Average, With <6, 6-10, >=6, 10-14, and >14 Doses Per Month
Description: The calculation of baseline and post-baseline mean BP (either systolic or diastolic) for each month (30-day period) is the average of all valid T-SMBP measurements. The subgrouping of the ITT population was created and examined to demonstrate the robustness of the results for the primary analysis. Descriptive statistics were calculated for baseline, month 6, and change from baseline to month 6. LSMeans and corresponding confidence intervals (CIs) were based on MMRM analysis. LSMeans and CIs were not calculated for the 10-14 and the >14 doses/month groups due to lack of convergence.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sumatriptan/Naproxen
Number analyzed (Participants) | 122
mmHg
  Systolic,<6 doses per month | -1.6 [-3.1 to 0.0]
  Systolic, 6-10 doses per month | -4.6 [-7.4 to -1.8]
  Systolic, >=6 doses per month | -4.3 [-7.1 to -1.6]
  Diastolic,<6 doses per month | -1.0 [-2.2 to 0.3]
  Diastolic, 6-10 doses per month | -3.7 [-7.1 to -0.4]
  Diastolic, >=6 doses per month | -3.5 [-6.3 to -0.7]

8. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure at Month 6 for Sumatriptan/Naproxen for the ITT Subpopulation of Participants Treating With <30 Total Doses, 30-60 Total Doses, >=30, 60-90 Total Doses, and >90 Total Doses
Description: The calculation of baseline and post-baseline mean BP (either systolic or diastolic) for each month (30-day period) is the average of all valid T-SMBP measurements. The subgrouping of the ITT population was created and examined to demonstrate the robustness of the results for the primary analysis. Descriptive statistics were calculated for baseline, month 6, and change from baseline to month 6. LSMeans and corresponding confidence intervals (CIs) were based on MMRM analysis. LSMeans and CIs were not calculated for the 60-90 and the >90 total dose groups due to lack of convergence.
Time Frame: Baseline and Month 6
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Sumatriptan/Naproxen
Number analyzed (Participants) | 122
mmHg
  Systolic, <30 total doses | -1.2 [-2.9 to 0.4]
  Systolic, 30-60 total doses | -3.4 [-6.0 to -0.7]
  Systolic, >=30 total doses | -3.7 [-6.0 to -1.4]
  Diastolic, <30 total doses | -0.6 [-2.0 to 0.7]
  Diastolic, 30-60 total doses | -3.3 [-5.8 to -0.8]
  Diastolic, >=30 total doses | -3.6 [-5.7 to -1.4]

9. Secondary Outcome: Number of Participants With an Increase of >=5 mmHg From the Baseline Systolic Blood Pressure for the Average of Any Given Two-day Consecutive Collection of Blood Pressure Measurements
Description: The number of participants with an increase of >=5 mmHg from the baseline systolic blood pressure for the average of any given two-day consecutive collection of valid blood pressure measurements during the study were summarized. Valid blood pressure measurements were defined as follows: must be taken at least 24 hours following last dose of investigational product used to treat an individual migraine, must be taken no later than 96 hours after last dose of investigational product used to treat an individual migraine, must be taken prior to the onset of a subsequent individual migraine.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population. Only participants with valid blood pressure measurements were analyzed.
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 120 | 109 | 115
participants | 53 | 57 | 63
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.9 to 2.6]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.9 to 2.6]

10. Secondary Outcome: Number of Participants With an Increase of >=3 mmHg From the Baseline Diastolic Blood Pressure for the Average of Any Given Two-day Consecutive Collection of Blood Pressure Measurements
Description: The number of participants with an increase of >=3 mmHg from the baseline diastolic blood pressure for the average of any given two-day consecutive collection of valid blood pressure measurements during the study were summarized. Valid blood pressure measurements were defined as follows: must be taken at least 24 hours following last dose of investigational product used to treat an individual migraine, must be taken no later than 96 hours after last dose of investigational product used to treat an individual migraine, must be taken prior to the onset of a subsequent individual migraine.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population. Only participants with valid blood pressure measurements were analyzed.
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 120 | 109 | 115
participants | 72 | 65 | 77
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.7]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.7 to 2.2]

11. Secondary Outcome: Number of Participants With a Consecutive 2-day Average Systolic Blood Pressure of >=140 mmHg During the Study
Description: The number of participants with any valid two-day consecutive average systolic blood pressure measurement of >=140 mmHg was calculated. Valid blood pressure measurements were defined as follows: must be taken at least 24 hours following last dose of investigational product used to treat an individual migraine, must be taken no later than 96 hours after last dose of investigational product used to treat an individual migraine, must be taken prior to the onset of a subsequent individual migraine.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 122 | 112 | 118
participants | 2 | 2 | 3
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.1 to 13.6]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Odds Ratio (OR) = 2.8, 95% CI 2-sided [0.3 to 25.6]

12. Secondary Outcome: Number of Participants With a Consecutive 2-day Average Diastolic Blood Pressure of >=90 mmHg
Description: The number of participants with any valid two-day consecutive average diastolic blood pressure measurement of >=90 mmHg was calculated. Valid blood pressure measurements were defined as follows: must be taken at least 24 hours following last dose of investigational product used to treat an individual migraine, must be taken no later than 96 hours after last dose of investigational product used to treat an individual migraine, must be taken prior to the onset of a subsequent individual migraine.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 122 | 112 | 118
participants | 10 | 11 | 11
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.5 to 3.7]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.6 to 4.2]

13. Secondary Outcome: Time to the First Day With an Average Systolic Blood Pressure Increase of >=5 mmHg From the Baseline Systolic Blood Pressure
Description: Kaplan-Meier curves for the distribution of time to the first day with an average diastolic BP increase of >=3 mmHg from the baseline diastolic BP during each calendar day were calculated and graphed for each treatment group. Only valid BP measurements were included and were defined as follows: must be taken at least 24 hours following last dose of investigational product used to treat an individual migraine, must be taken no later than 96 hours after last dose of investigational product used to treat an individual migraine, must be taken prior to the onset of a subsequent individual migraine.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population. Only participants with valid blood pressure measurements were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 120 | 109 | 115
days | 42.5 [2 to 177] | 32.5 [3 to 118] | 18.5 [3 to 124]
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.84 to 1.54]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [1.01 to 1.83]

14. Secondary Outcome: Time to the First Day With an Average Diastolic Blood Pressure Increase of >=3 mmHg From the Baseline Diastolic Blood Pressure
Description: as for outcome 13
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population. Only participants with valid blood pressure measurements were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 120 | 109 | 115
days | 51 [2 to 140] | 50.5 [3 to 161] | 26 [3 to 124]
Statistical Analysis 1: Comparison: Sumatriptan/Naproxen vs Sumatriptan; Test type: Superiority or Other; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.65 to 1.21]
Statistical Analysis 2: Comparison: Sumatriptan/Naproxen vs Naproxen; Test type: Superiority or Other; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.88 to 1.60]

15. Secondary Outcome: Number of Participants Withdrawn From the Study Due to Blood Pressure Changes
Description: The number of participants withdrawn from the study due to protocol-defined blood pressure changes were summarized for each treatment group. Defined blood pressure changes included (1) monthly average BP ≥140 mmHg systolic or >=90 mmHg diastolic and confirmed in clinic, (2) monthly average BP increase of >=30 mmHg systolic or >=20 mmHg from in-clinic screening and confirmed in clinic, and (3) systolic >=140 mmHg or diastolic >=90 mmHg on consecutive clinic visits >=2 weeks apart.
Time Frame: Baseline to End of Study (6-month study duration)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Number analyzed (Participants) | 122 | 112 | 118
participants | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and adverse events (AEs) were recorded from the start of investigational product and until any follow-up contact
Description: SAEs and AEs were collected in the Safety Population, which is comprised of all participants who took at least one dose of investigational product. SAE term "abortion induced" was actually coded to surgical and medical procedures in the MedDRA dictionary; however, this organ system is not available in the current template drop-down list.
Arm/Group | Sumatriptan/Naproxen | Sumatriptan | Naproxen
Serious Adverse Events (participants affected / at risk) | 3/127 | 1/120 | 0/127
Other Adverse Events (participants affected / at risk) | 20/127 | 29/120 | 18/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sumatriptan/Naproxen (N=127) | Sumatriptan (N=120) | Naproxen (N=127)
Chest pain (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abortion induced (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sumatriptan/Naproxen (N=127) | Sumatriptan (N=120) | Naproxen (N=127)
Nasopharyngitis (Infections and infestations) | 4 | 6 | 5
Urinary tract infection (Infections and infestations) | 1 | 6 | 3
Sinusitis (Infections and infestations) | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 1
Dizziness (Nervous system disorders) | 5 | 5 | 1
Somnolence (Nervous system disorders) | 2 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 1
Seasonal allergy (Immune system disorders) | 3 | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.